CLINICAL TRIAL: NCT05235542
Title: A Phase Ib/II Study of AK104#PD-1 / CTLA-4 Bispecific Antibody# and AK117#Anti-CD47 Antibody# in Combination With or Without Chemotherapy in Advanced Malignant Tumors
Brief Title: A Phase Ib/II Study of AK104 and AK117 in Combination With or Without Chemotherapy in Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK117-204
Record Dates: First submitted 2022-01-25; First posted 2022-02-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Advanced Malignant Tumors
MeSH Terms: interventions — Capecitabine; Oxaliplatin; Cisplatin; Paclitaxel; Irinotecan; Docetaxel; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase Ib#Dosage regimen 1# (Experimental): Subjects receive AK104 plus AK117 every 3- week cycle (Q3W) until progression
  Interventions: Drug: AK104; Drug: AK117
- Phase Ib#Dosage regimen 2# (Experimental): Subjects receive AK104 plus AK117 every 6- week cycle (Q6W) until progression
  Interventions: Drug: AK104; Drug: AK117
- Phase II#Cohort 1# (Experimental): Gastric Cancer or Gastroesophageal Junction Cancer: AK104 + XELOX (Oxaliplatin + Capecitabine)+AK117 every 3- week cycle (Q3W) until progression
  Interventions: Drug: AK104; Drug: AK117; Drug: Capecitabine tablets; Drug: Oxaliplatin
- Phase II#Cohort 2# (Experimental): Esophageal squamous cell cancer: AK104 + 5-FU/Paclitaxel+Cisplatin± AK117 every 3- week cycle (Q3W) until progression
  Interventions: Drug: AK104; Drug: AK117; Drug: Cisplatin; Drug: Paclitaxel; Drug: 5-FU
- Phase II#Cohort 3# (Experimental): Gastric Cancer or Gastroesophageal Junction Cancer or Esophageal squamous cell cancer: AK117 +Paclitaxel/Docetaxel/Irinotecan every 3- or 4- week cycle (Q3W or Q4W) until progression
  Interventions: Drug: AK117; Drug: Paclitaxel; Drug: Irinotecan; Drug: Docetaxel

INTERVENTIONS:
Drug: AK104 — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 1#; Phase II#Cohort 2#; Phase Ib#Dosage regimen 1#; Phase Ib#Dosage regimen 2#
Drug: AK117 — IV infusion,Specified dose on specified days
Drug: Capecitabine tablets — Oral,Specified dose on specified days
  Arms: Phase II#Cohort 1#
Drug: Oxaliplatin — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 1#
Drug: Cisplatin — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 2#
Drug: Paclitaxel — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 2#; Phase II#Cohort 3#
Drug: Irinotecan — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 3#
Drug: Docetaxel — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 3#
Drug: 5-FU — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 2#

SUMMARY:
Phase Ib/II open label, multicenter study to evaluate the efficacy and safety of AK104 (anti-PD-1 and CTLA-4 bispecific antibody) and AK117#AntiCD47 Antibody# combined with or without chemotherapy in advanced malignant tumors

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old.
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Have a life expectancy of at least 3 months.
4. Phase Ib: Histologically or cytologically confirmed advanced solid tumor.
5. Phase II: Has histologically confirmed diagnosis of unresectable locally advanced,recurrent or metastatic gastric or GEJ adenocarcinoma or Esophageal squamous cell carcinoma.
6. Have at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator.
7. Has adequate organ function.

Exclusion Criteria:

1. Undergone major surgery within 30 days prior to the first dose of study treatment.
2. Active central nervous system (CNS) metastases.
3. History of active autoimmune disease that has required systemic treatment in the past 2 years (i.e.,corticosteroids or immunosuppressive drugs).
4. Active Hepatitis B or Hepatitis C.
5. Received previous immunotherapy, including immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy and other treatments targeting the mechanism of tumor immunity.
6. History of severe bleeding tendency or coagulation disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Adverse Events (AEs) | Up to approximately 2 years
Objective Response Rate (ORR) | Up to approximately 2 years

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
Duration of Response (DoR) | Up to approximately 2 years
Time to response (TTR) | Up to approximately 2 years
Progression free survival (PFS) | Up to approximately 2 years
Overall survival (OS) | Up to approximately 2 years
Maximum observed concentration (Cmax) of AK117 and AK104 | From first dose of study drug to last dose of of study drug
  The endpoints for assessment of PK include serum concentrations of AK117 and AK104 at different timepoints after study drug administration.
Minimum observed concentration (Cmin) of AK117 and AK104 at steady state | From first dose of study drug to last dose of of study drug
  The endpoints for assessment of PK include serum concentrations of AK117 and AK104 at different timepoints after study drug administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of study drug through 30 days after last dose of study drug
  The immunogenicity of AK117 and AK104 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Wang, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Shanghai Renji Hospital, Shanghai, China